CLINICAL TRIAL: NCT03398135
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled 52-Week Maintenance and an Open-Label Extension Study of the Efficacy and Safety of Risankizumab in Subjects With Ulcerative Colitis
Brief Title: A Study to Assess the Efficacy and Safety of Risankizumab in Participants With Ulcerative Colitis
Acronym: COMMAND
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M16-066; 2023-506994-36-00 (Other: EU CT)
Record Dates: First submitted 2018-01-08; First posted 2018-01-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis (UC)
Keywords: ABBV-066; BI 655066
MeSH Terms: conditions — Colitis, Ulcerative | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Substudy 1: Double-blind Placebo (Placebo Comparator): Participants randomized to receive placebo for risankizumab administered by subcutaneous (SC) injection.
  Interventions: Drug: placebo for risankizumab
- Substudy 1: Double-blind Risankizumab Dose 1 (Experimental): Participants randomized to receive risankizumab dose 1 administered by subcutaneous (SC) injection.
  Interventions: Drug: risankizumab
- Substudy 1: Double-blind Risankizumab Dose 2 (Experimental): Participants randomized to receive risankizumab dose 2 administered by subcutaneous (SC) injection.
  Interventions: Drug: risankizumab
- Substudy 2: Open-label (OL) Clinical Assessment Risankizumab (Experimental): Participants randomized to receive risankizumab dose 1 administered by subcutaneous (SC) injection.
  Interventions: Drug: risankizumab
- Substudy 2: OL Therapeutic Drug Monitoring Risankizumab (Experimental): Participants randomized to receive risankizumab dose 1 administered by subcutaneous (SC) injection.
  Interventions: Drug: risankizumab
- Substudy 3: OL Extension Risankizumab (Experimental): Participants who completed Sub-study 1 or 2 receive open-label risankizumab in Sub-study 3.
  Interventions: Drug: risankizumab
- OL Continuous Treatment Extension - Dose 1 (Experimental): Participants who complete Sub-study 3 and continue to tolerate and derive benefit from receiving risankizumab, will continue to receive risankizumab based on their assignment during Sub-study 3. Participants completing Sub-study 3 without receiving risankizumab rescue therapy in any sub-study will receive risankizumab Dose 1 administered by subcutaneous (SC) injection.
  Interventions: Drug: risankizumab
- OL Continuous Treatment Extension - Dose 2 (Experimental): Participants who complete Sub-study 3 and continue to tolerate and derive benefit from receiving risankizumab, will continue to receive risankizumab based on their assignment during Sub-study 3. Participants completing Sub-study 3 and received risankizumab rescue therapy in any sub-study will receive risankizumab Dose 2 administered by subcutaneous (SC) injection.
  Interventions: Drug: risankizumab

INTERVENTIONS:
Drug: risankizumab — subcutaneous (SC) injection
  Other Names: ABBV-066; BI 655066; SKYRIZI
  Arms: OL Continuous Treatment Extension - Dose 1; OL Continuous Treatment Extension - Dose 2; Substudy 1: Double-blind Risankizumab Dose 1; Substudy 1: Double-blind Risankizumab Dose 2; Substudy 2: OL Therapeutic Drug Monitoring Risankizumab; Substudy 2: Open-label (OL) Clinical Assessment Risankizumab; Substudy 3: OL Extension Risankizumab
Drug: placebo for risankizumab — subcutaneous (SC) injection
  Arms: Substudy 1: Double-blind Placebo

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of risankizumab in participants with ulcerative colitis (UC) in participants who responded to induction treatment with risankizumab in a prior AbbVie study of risankizumab in UC.

This study consists of three sub-studies and a Continuous Treatment Extension (CTE): Substudy 1 is a 52-week, randomized, double-blind, placebo-controlled maintenance study; Substudy 2 is 52-week, randomized, exploratory maintenance study; and Substudy 3 is an open-label long-term extension study for participants who completed Substudy 1 or 2, or participants who responded to induction treatment in Study M16-067 with no final endoscopy due to the Covid-19 pandemic or due to the geopolitical conflict in Ukraine and surrounding impacted regions. The CTE is an open-label extension for Substudy 3 completers to ensure continuous treatment with risankizumab until such time that risankizumab becomes commercially available and/or the subject can access treatment locally.

ELIGIBILITY:
Inclusion Criteria:

- Participants who have completed Study M16-067 and have achieved clinical response as defined in the protocol.

Exclusion Criteria:

* Participants who have a known hypersensitivity to risankizumab or the excipients of any of the study drugs or the ingredients of chinese hamster ovary (CHO) or had an adverse event (AE) during Studies M16-067 that in the Investigator's judgment makes the participant unsuitable for this study.
* Participant is considered by the Investigator, for any reason, to be an unsuitable candidate for the study.
* Participant is not in compliance with prior and concomitant medication requirements throughout Studies M16-067.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1242 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Sub-Study 1: Percentage of Participants Achieving Clinical Remission per Adapted Mayo Score | Week 52
  Clinical remission per Adapted Mayo Score.
Percentage of Participants with Adverse Events (AE) | Up to Week 300
  An Adverse Event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Sub-Study 1: Percentage of Participants Achieving Endoscopic Improvement | Week 52
  Endoscopic improvement per endoscopy subscore.
Sub-Study 1: Percentage of Participants Achieving Histologic-Endoscopic Mucosal Improvement | Week 52
  Percentage of participants achieving histologic-endoscopic mucosal improvement.
Sub-Study 1: Percentage of Participants Achieving Endoscopic Remission | Week 52
  Endoscopic remission per endoscopy subscore.
Sub-Study 1: Percentage of Participants with Clinical Remission per Adapted Mayo Score in Participants with no Corticosteroid Use for 90 days | Week 52
  Clinical remission per Adapted Mayo Score.
Sub-Study 1: Percentage of Participants with Clinical Remission per Adapted Mayo Score in Participants with a Clinical Remission at Week 0 | Week 52
  Clinical remission per Adapted Mayo Score.
Sub-Study 1: Percentage of Participants Achieving No Bowel Urgency | Week 52
  Percentage of participants achieving no bowel urgency.
Sub-Study 1: Percentage of Participants Achieving No Abdominal Pain | Week 52
  Percentage of participants achieving no abdominal pain.
Sub-Study 1: Percentage of Participants Achieving Histologic-Endoscopic Mucosal Remission | Week 52
  Percentage of participants achieving histologic-endoscopic mucosal remission per endoscopy subscore.
Sub-Study 1: Percentage of Participants Achieving Endoscopic Improvement in Participants with Endoscopic Improvement at Week 0 | Week 52
  Endoscopic improvement per endoscopy subscore.
Sub-Study 1: Percentage of Participants Achieving Clinical Response per Adapted Mayo Score | Week 52
  Clinical response per Adapted Mayo Score.
Sub-Study 1: Change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) | Week 0 to Week 52
  The FACIT-Fatigue is a validated tool that measures an individual's level of fatigue during their usual daily activities over the past week.
Sub-Study 1: Change in Inflammatory Bowel Disease Questionnaire (IBDQ) | Baseline (Week 0) to Week 52
  The IBDQ is used to assess the quality of life of patients with inflammatory bowel disease.
Sub-Study 1: Percentage of Participants Achieving No Nocturnal Bowel Movements | Week 52
  Percentage of participants achieving no nocturnal bowel movements.
Sub-Study 1: Percentage of Participants Achieving No Tenesmus | Week 52
  Percentage of participants achieving no tenesmus.
Sub-Study 1: Change in Number of Fecal Incontinence Episodes per Week | Baseline (Week 0) to Week 52
  Change in number of fecal incontinence episodes per week.
Sub-Study 1: Change in Number of Days per Week with Sleep Interrupted due to UC Symptoms | Baseline (Week 0) to Week 52
  Change in number of days per week with sleep interrupted due to UC symptoms.
Sub-Study 1: Percentage of Participants with Exposure Adjusted Occurrence of Ulcerative Colitis (UC) Related Hospitalization | Through Week 52
  Participants with an exposure adjusted occurrence of UC event that results in admission to the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (426):
- United States (78):
  - Southern California Res. Ctr. /ID# 169659, Coronado, California
  - Hoag Memorial Hosp Presbyterian /ID# 218347, Irvine, California
  - UC San Diego Health System /ID# 160430, La Jolla, California
  - United Medical Doctors /ID# 158574, Los Alamitos, California
  - Cedars-Sinai Medical Center /ID# 163848, Los Angeles, California
  - Gastrointestinal Biosciences Clinical Trials, LLC /ID# 200934, Los Angeles, California
  - UCSF Medical Center - Mount Zion /ID# 201209, San Francisco, California
  - Peak Gastroenterology Associates, PC /ID# 165838, Colorado Springs, Colorado
  - Rocky Mountain Pediatric Gastroenterology /ID# 207173, Lone Tree, Colorado
  - Duplicate_Medical Research Center of CT /ID# 160287, Hamden, Connecticut
  - Yale Univ Digestive Diseases /ID# 213265, New Haven, Connecticut
  - South Lake Pain Institute, Inc /ID# 162859, Clermont, Florida
  - Ctr for Advanced Gastroenterol /ID# 202820, Maitland, Florida
  - University of Miami /ID# 160456, Miami, Florida
  - Coral Research Clinic /ID# 158608, Miami, Florida
  - South Florida Research Ph I-IV, Inc. /ID# 161844, Miami, Florida
  - Gastroenterology Group Naples /ID# 165210, Naples, Florida
  - Advanced Research Institute, Inc /ID# 161945, New Port Richey, Florida
  - Advent Health /ID# 160393, Orlando, Florida
  - Endoscopic Research, Inc. /ID# 206709, Orlando, Florida
  - Omega Research Group /ID# 203105, Orlando, Florida
  - Duplicate_Lenus Research & Medical Group /ID# 169727, Sweetwater, Florida
  - Clinical Research Trials of Florida, Inc. /ID# 201794, Tampa, Florida
  - Duplicate_AdventHealth Tampa /ID# 170482, Tampa, Florida
  - Gastroenterology Associates of Central Georgia, LLC /ID# 160513, Macon, Georgia
  - The University of Chicago Medical Center /ID# 160511, Chicago, Illinois
  - DM Clinical Research/Southwest /ID# 165009, Oak Lawn, Illinois
  - Indiana University /ID# 167250, Indianapolis, Indiana
  - Univ Kansas Med Ctr /ID# 226601, Kansas City, Kansas
  - Cotton O'Neil Clinical Research Center, Digestive Health /ID# 160367, Topeka, Kansas
  - Duplicate_Robley Rex VA Medical Center /ID# 218647, Louisville, Kentucky
  - Houma Digestive Health Special /ID# 158377, Houma, Louisiana
  - Delricht Research /ID# 206817, New Orleans, Louisiana
  - Nola Research Works, LLC /ID# 161356, New Orleans, Louisiana
  - Louisiana Research Center, LLC /ID# 201205, Shreveport, Louisiana
  - Massachusetts General Hospital - Crohn's and Colitis Center /ID# 164257, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 159430, Ann Arbor, Michigan
  - Clin Res Inst of Michigan, LLC /ID# 160300, Chesterfield, Michigan
  - Mayo Clinic - Rochester /ID# 200455, Rochester, Minnesota
  - Quality Clinical Research Inc. /ID# 167312, Omaha, Nebraska
  - Weill Cornell Medicine /ID# 165884, New York, New York
  - Columbia Univ Medical Center /ID# 161929, New York, New York
  - Lenox Hill Hospital /ID# 168469, New York, New York
  - Manhattan Clinical Research, LLC /ID# 211803, New York, New York
  - Duplicate_DiGiovanna Institute for Medical Education & Research /ID# 171128, North Massapequa, New York
  - Duplicate_University of Rochester Medical Center /ID# 161660, Rochester, New York
  - Atrium Health Carolinas Medical Center /ID# 158543, Charlotte, North Carolina
  - Plains Clinical Research Center, LLC /ID# 169729, Fargo, North Dakota
  - Cleveland Clinic Main Campus /ID# 209235, Cleveland, Ohio
  - The Ohio State University /ID# 164713, Columbus, Ohio
  - Optimed Research, Ltd. /ID# 167112, Columbus, Ohio
  - Great Lakes Gastroenterology Research, LLC /ID# 201778, Mentor, Ohio
  - ProMedica Physicians Digestive Healthcare /ID# 215622, Sylvania, Ohio
  - Digestive Disease Specialists /ID# 170777, Oklahoma City, Oklahoma
  - Adult Gastroenterology Associates - Gen 1 Research /ID# 208873, Tulsa, Oklahoma
  - Penn State Milton S. Hershey Medical Center /ID# 230474, Hershey, Pennsylvania
  - University of Pennsylvania /ID# 166262, Philadelphia, Pennsylvania
  - Digestive Disease Associates, LTD - Wyomissing /ID# 232406, Wyomissing, Pennsylvania
  - Gastroenterology Associates, P.A. of Greenville /ID# 160457, Greenville, South Carolina
  - Gastro One /ID# 160373, Cordova, Tennessee
  - Duplicate_East Tennessee Research Institute /ID# 168744, Johnson City, Tennessee
  - Vanderbilt University Medical Center /ID# 160567, Nashville, Tennessee
  - Inquest Clinical Research /ID# 165686, Baytown, Texas
  - Texas Digestive Disease Consultants /ID# 209951, Cedar Park, Texas
  - GI Alliance /ID# 209799, Cedar Park, Texas
  - Digestive Health Associates of Texas (DHAT) Research Institute - Garland /ID# 158235, Garland, Texas
  - Vilo Research Group Inc /ID# 207657, Houston, Texas
  - Baylor College of Medicine /ID# 158230, Houston, Texas
  - Centex Studies, Inc. - Houston /ID# 201221, Houston, Texas
  - Duplicate_Caprock Gastro Research, LLC /ID# 215433, Lubbock, Texas
  - Clinical Associates in Research Therapeutics of America, LLC /ID# 161364, San Antonio, Texas
  - Southern Star Research Institute, LLC /ID# 168774, San Antonio, Texas
  - Baylor Scott & White Center for Diagnostic Medicine /ID# 204132, Temple, Texas
  - Tyler Research Institute, LLC /ID# 166799, Tyler, Texas
  - Gastro Health & Nutrition - Victoria /ID# 164308, Victoria, Texas
  - Advanced Research Institute /ID# 160465, Ogden, Utah
  - Gastroenterology Consultants of Southwest Virginia /ID# 218142, Roanoke, Virginia
  - Virginia Mason Hospital & Medical Center /ID# 160432, Seattle, Washington
- Argentina (5):
  - Cemic /Id# 167805, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Gedyt /ID# 243424, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Hospital Provincial del Centenario /ID# 170896, Rosario, Santa Fe Province
  - Sanatorio 9 de Julio /ID# 167803, San Miguel de Tucumán, Tucumán Province
  - Hospital Privado Universitario - Hospital Privado Centro Medico de Cordoba S.A. /ID# 167802, Córdoba
- Austria (5):
  - Duplicate_Universitaetsklinikum St.Poelten /ID# 169049, Sankt Pölten, Lower Austria
  - Duplicate_Medizinische Universitaet Graz /ID# 169052, Graz, Styria
  - Ordensklinikum Linz GmbH Barmherzige Schwestern /ID# 216043, Linz, Upper Austria
  - Medizinische Universitaet Wien /ID# 169051, Vienna, Vienna
  - Landeskrankenhaus Salzburg-Universitaetsklinikum der PMU (LKH) /ID# 200686, Salzburg
- Belgium (8):
  - Imelda Ziekenhuis /ID# 211101, Bonheiden, Antwerpen
  - Universite Libre de Bruxelles - Hopital Erasme /ID# 200256, Anderlecht, Brussels Capital
  - Cliniques Universitaires UCL Saint-Luc /ID# 200260, Brussels, Brussels Capital
  - Groupe Sante CHC - Clinique du MontLegia /ID# 200255, Liège, Liege
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant /ID# 200259, Yvoir, Namur
  - Universitair Ziekenhuis Leuven /ID# 170829, Leuven, Vlaams-Brabant
  - AZ-Delta /ID# 200258, Roeselare, West-Vlaanderen
  - CHU de Liege /ID# 200257, Liège
- Brazil (7):
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva /ID# 157683, Goiânia, Goiás
  - Faculdade de Medicina do ABC /ID# 163993, Santo André, La Spezia
  - Hospital Nossa Senhora das Graças /ID# 157677, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre /ID# 157670, Porto Alegre, Rio Grande do Sul
  - Upeclin Fmb - Unesp /Id# 157691, Botucatu, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto /ID# 157668, Ribeirão Preto, São Paulo
  - Kaiser Clinica e Hospital Dia /ID# 157686, São José do Rio Preto, São Paulo
- Bulgaria (5):
  - Hospital Tsaritsa Yoanna /ID# 209978, Sofiya, Sofia
  - Umbal Kaspela /ID# 200795, Plovdiv
  - MHAT Hadzhi Dimitar /ID# 207947, Sliven
  - Duplicate_Second MHAT Sofia /ID# 200794, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 210798, Sofia
- Canada (11):
  - Duplicate_University of Calgary /ID# 169125, Calgary, Alberta
  - Allen Whey Khye Lim Professional Corporation /ID# 169770, Edmonton, Alberta
  - Covenant Health /ID# 169128, Edmonton, Alberta
  - Fraser Clinical Trials Inc /ID# 169116, New Westminster, British Columbia
  - Percuro Clinical Research, Ltd /ID# 169123, Victoria, British Columbia
  - London Health Sciences Center- University Hospital /ID# 169117, London, Ontario
  - Scott Shulman Medicine Professional Corporation /ID# 169127, North Bay, Ontario
  - Toronto Digestive Disease Associates /ID# 169120, Vaughan, Ontario
  - Hotel Dieu de Levis /ID# 214379, Lévis, Quebec
  - CIUSSS de l'est de l'Ile-de-Montreal - Hopital Maisonneuve-Rosemont /ID# 169122, Montreal, Quebec
  - Montreal General Hospital- McGill University Health Center /ID# 169118, Montreal, Quebec
- Chile (4):
  - Hospital Guillermo Grant Benavente de Concepción /ID# 210762, Concepción, Bio-Bio
  - Hospital Las Higueras /ID# 167094, Talcahuano, Bio-Bio
  - Duplicate_Servicio de Salud Araucanía Norte Hospital Victoria /ID# 213152, Victoria, Región de la Araucanía
  - Complejo Asistencial Dr. Sotero del Rio /ID# 169386, Santiago, Santiago Metropolitan
- China (25):
  - The First Affiliated Hospital of Anhui Medical University /ID# 211227, Hefei, Anhui
  - Beijing Friendship Hospital /ID# 211061, Beijing, Beijing Municipality
  - The Sixth Affiliated Hospital of Sun Yat-sen University /ID# 211229, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University /ID# 213019, Shijiazhuang, Hebei
  - Tongji Hospital Tongji Medical College of HUST /ID# 211069, Wuhan, Hubei
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Sc /ID# 211070, Wuhan, Hubei
  - Renmin Hospital of Wuhan University /ID# 212867, Wuhan, Hubei
  - The Second Xiangya Hospital Of Central South University /ID# 211196, Changsha, Hunan
  - Huai'an First People's Hospital /ID# 239197, Huaian, Jiangsu
  - Nanjing Drum Tower Hospital /ID# 227438, Nanjing, Jiangsu
  - Jiangsu Province Hospital /ID# 211234, Nanjing, Jiangsu
  - Wuxi People's Hospital /ID# 218797, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 212182, Nanchang, Jiangxi
  - The First Hospital of Jilin University /ID# 212277, Changchun, Jilin
  - Shengjing Hospital of China Medical University /ID# 211643, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University /ID# 213912, Yinchuan, Ningxia
  - Xijing Hospital /ID# 210708, Xi'an, Shaanxi
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 210960, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine /ID# 211230, Shanghai, Shanghai Municipality
  - Shanghai East Hospital /ID# 218796, Shanghai, Shanghai Municipality
  - Shanghai General Hospital /ID# 226652, Shanghai, Shanghai Municipality
  - Tangdu Hospital of The Fourth Military Medical University, PLA /ID# 215505, Xi’an, Shanxi
  - West China Hospital, Sichuan University /ID# 211275, Chengdu, Sichuan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine /ID# 211024, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital,Meical School Zhejiang University /ID# 211062, Hangzhou, Zhejiang
- Colombia (3):
  - Fundación Hospitalaria San Vicente de Paul /ID# 171488, Medellín, Antioquia
  - Coorp Hosp Juan Ciudad Sede Hospital Universitario Mayor Mederi /ID# 158736, Bogota DC, Cundinamarca
  - Imat Oncomedica /ID# 207041, Montería, Departamento de Córdoba
- Croatia (5):
  - Clinical Hospital Dubrava /ID# 157598, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 157594, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 201915, Zagreb, City of Zagreb
  - Poliklinika Borzan d.o.o. /ID# 157595, Osijek, County of Osijek-Baranja
  - Klinicki Bolnicki Centar (KBC) Split /ID# 157596, Split, Split-Dalmatia County
- Czechia (5):
  - Duplicate_Fakultni nemocnice u sv. Anny v Brne /ID# 239158, Brno, Brno-mesto
  - Fakultni Nemocnice Ostrava /ID# 225568, Ostrava, Ostrava-mesto
  - SurGal Clinic /ID# 252300, Brno, South Moravian
  - Nemocnice Ceske Budejovice a.s. /ID# 225228, České Budějovice
  - Hepato-Gastroenterologie HK, s.r.o. /ID# 163389, Hradec Králové
- Denmark (4):
  - Bispebjerg and Frederiksberg Hospital /ID# 208953, Copenhagen NV, Capital Region
  - Kobenhavns Universitet - Hvidovre Hospital (HH) /ID# 205093, Hvidovre, Capital Region
  - Duplicate_Sjællands Universitetshospital /ID# 200073, Roskilde, Region Sjælland
  - Duplicate_Odense Universitets Hospital /ID# 209502, Odense C, Region Syddanmark
- Egypt (5):
  - Alexandria University /ID# 226795, Alexandria, Alexandria Governorate
  - Alexandria University /ID# 226796, Alexandria, Alexandria Governorate
  - National Liver Institute /ID# 171042, Menoufiya, Monufia Governorate
  - Duplicate_Clinical Research Center, Faculty of Medicine, Alexandria university. /ID# 201824, Alexandria
  - Air Force Specialized Hospital /ID# 170984, Cairo
- France (10):
  - Chu de Nice-Hopital Larchet Ii /Id# 207881, Nice, Alpes-Maritimes
  - APHM - Hopital Nord /ID# 225826, Marseille, Bouches-du-Rhone
  - CHU Montpellier - Hopital Saint Eloi /ID# 223781, Montpellier, Herault
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois /ID# 207877, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Centre Hospitalier Universitaire de Bordeaux /ID# 207883, Pessac, Nouvelle-Aquitaine
  - Duplicate_CHU de SAINT ETIENNE - Hopital Nord /ID# 207882, Saint Priest EN Jarez, Pays de la Loire Region
  - Duplicate_CHU Amiens-Picardie Site Sud /ID# 207880, Amiens, Somme
  - Clinique Jules Verne /ID# 240977, Nantes
  - Hopital Beaujon /ID# 207876, Clichy, Île-de-France Region
  - Centre Medico Chirurgical Ambroise Pare Hartmann /ID# 249861, Neuilly-sur-Seine, Île-de-France Region
- Germany (20):
  - Universitaetsklinikum Freiburg /ID# 162038, Freiburg im Breisgau, Baden-Wurttemberg
  - Praxis fuer Gastroenterologie /ID# 166154, Heidelberg, Baden-Wurttemberg
  - Universitatsklinikum Mannheim /ID# 162039, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 164994, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 159373, Erlangen, Bavaria
  - Duplicate_LMU Klinikum Campus Grosshadern /ID# 210484, Munich, Bavaria
  - Duplicate_Agaplesion Markus Krankenhaus /ID# 159375, Frankfurt am Main, Hesse
  - Gastroenterologie Opernstrasse Private Practice - Dr. Falk & Krause & Kuhn /ID# 163690, Kassel, Hesse
  - Klinikum Lueneburg /ID# 163692, Lüneburg, Lower Saxony
  - Universitaetsklinikum Koeln /ID# 164993, Cologne, North Rhine-Westphalia
  - Praxiszentrum fuer Gastroenterologie /ID# 219072, Grevenbroich, North Rhine-Westphalia
  - Gastroenterologische Gemeinschaftspraxis Minden /ID# 162037, Minden, North Rhine-Westphalia
  - Eugastro /ID# 219071, Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 159379, Kiel, Schleswig-Holstein
  - Gastroenterologische Spezialpraxis am Wittenbergplatz /ID# 219146, Berlin
  - MVZ fuer Gastroenterlogie am Bayerischen Platz /ID# 159380, Berlin
  - Charite Universitaetsklinikum Berlin - Campus Benjamin Franklin /ID# 210508, Berlin
  - DRK Kliniken Berlin Westend /ID# 166155, Berlin
  - Stadtisches Klinikum Braunschweig /ID# 163694, Braunschweig
  - Universitaetsklinikum Regensburg /ID# 163693, Regensburg
- Greece (8):
  - General Hospital of Athens Ippokratio /ID# 229190, Athens, Attica
  - General Hospital of Athens Laiko /ID# 206438, Athens, Attica
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 170910, Athens, Attica
  - General Hospital of Nikaia-Piraeus "Agios Panteleimon" /ID# 165313, Nikaia, Attica
  - Tzaneio general hospital of Piraeus /ID# 206437, Piraeus, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 165327, Heraklion, Crete
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 217479, Athens
  - Theageneio Anticancer Hospital /ID# 165329, Thessaloniki
- Israel (6):
  - Shaare Zedek Medical Center /ID# 163543, Jerusalem, Jerusalem
  - Hadassah Medical Center-Hebrew University /ID# 171092, Jerusalem, Jerusalem
  - Soroka University Medical Center /ID# 171093, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 211279, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus /ID# 171096, Haifa
  - Rabin Medical Center. /ID# 167402, Petah Tikva
- Italy (15):
  - Ospedale San Martino /ID# 164030, Genoa, Genova
  - IRCCS Istituto Clinico Humanitas /ID# 155626, Rozzano, Lombardy
  - ASST Fatebenefratelli Sacco /ID# 155623, Milan, Milano
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 170959, Milan, Milano
  - ASST Rhodense/Presidio Ospedaliero di Rho /ID# 211450, Rho, Milano
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 158020, Rome, Roma
  - Azienda Ospedaliera San Camillo Forlanini /ID# 155628, Rome, Roma
  - Duplicate_Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 171223, Rome, Roma
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 164029, Negrar, Verona
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 155627, Bologna
  - Ospedale Cannizzaro /ID# 164039, Catania
  - Azienda Ospedaliero-Universitaria Renato Dulbecco /ID# 200124, Catanzaro
  - Azienda Ospedaliero-Universitaria di Modena /ID# 201818, Modena
  - Fondazione Policlinico Universitario Campus Bio-Medico /ID# 163994, Roma
  - UOC Medicina Interna e Gastroe /ID# 155624, Rome
- Japan (61):
  - Aichi Medical University Hospital /ID# 164227, Nagakute, Aichi-ken
  - Daido Clinic - Nagoya /ID# 211478, Nagoya, Aichi-ken
  - Duplicate_Nagoya University Hospital /ID# 164230, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 164229, Nagoya, Aichi-ken
  - Fujita Health University Hospital /ID# 164313, Toyoake, Aichi-ken
  - National Hospital Organization Hirosaki General Medical Center /ID# 164216, Hirosaki-shi, Aomori
  - Tokatsu Tsujinaka Hospital /ID# 164310, Abiko-shi, Chiba
  - Chiba University Hospital /ID# 209633, Chiba, Chiba
  - Tsujinaka Hospital - Kashiwanoha /ID# 225968, Kashiwa-shi, Chiba
  - Toho University Sakura Medical Center /ID# 164219, Sakura-shi, Chiba
  - Fukuoka University Chikushi Hospital /ID# 209056, Chikushino-shi, Fukuoka
  - Saiseikai Fukuoka Genaral Hospital /ID# 225640, Fukuoka, Fukuoka
  - Fukuoka University Hospital /ID# 226723, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 164237, Kurume-shi, Fukuoka
  - Gifu University Hospital /ID# 208490, Gifu, Gifu
  - Ogaki Municipal Hospital /ID# 226009, Ogaki-shi, Gifu
  - National Hospital Organization Takasaki General Medical Center /ID# 164312, Takasaki-shi, Gunma
  - National Hospital Organization Fukuyama Medical Center /ID# 164315, Fukuyama-shi, Hiroshima
  - Hiroshima University Hospital /ID# 164240, Hiroshima, Hiroshima
  - Duplicate_Asahikawa Medical University Hospital /ID# 164324, Asahikawa-shi, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 164215, Sapporo, Hokkaido
  - Sapporo Medical University Hospital /ID# 164278, Sapporo, Hokkaido
  - Sapporo IBD Clinic /ID# 225967, Sapporo, Hokkaido
  - Sapporo Higashi Tokushukai Hospital /ID# 208493, Sapporo, Hokkaido
  - Aoyama Clinic /ID# 164236, Kobe, Hyōgo
  - Hyogo Medical University Hospital /ID# 164238, Nishinomiya-shi, Hyōgo
  - Kanazawa University Hospital /ID# 169221, Kanazawa, Ishikawa-ken
  - Sameshima Hospital /ID# 211182, Kagoshima, Kagoshima-ken
  - Tokai University Hospital /ID# 209207, Isehara, Kanagawa
  - Gokeikai Ofuna Chuo Hospital /ID# 169296, Kamakura-shi, Kanagawa
  - St Marianna University School Of Medicine /ID# 226730, Kawasaki-shi, Kanagawa
  - Kitasato University Hospital /ID# 169223, Sagamihara-shi, Kanagawa
  - Matsushima Hospital /ID# 254448, Yokohama, Kanagawa
  - Colo-proctology Center Matsushima Clinic /ID# 225915, Yokohama, Kanagawa
  - SHOWA Medical University Fujigaoka Hospital /ID# 209606, Yokohama, Kanagawa
  - Mie University Hospital /ID# 203635, Tsu, Mie-ken
  - Yokkaichi Hazu Medical Center /ID# 164316, Yokkaichi-shi, Mie-ken
  - Tohoku University Hospital /ID# 164276, Sendai, Miyagi
  - Duplicate_Nagasaki University Hospital /ID# 205326, Nagasaki, Nagasaki
  - Nara Medical University Hospital /ID# 169222, Kashihara-shi, Nara
  - Kinshukai Infusion Clinic /ID# 226992, Osaka, Osaka
  - Osaka Medical and Pharmaceutical University Hospital /ID# 226036, Takatsuki-shi, Osaka
  - Saga University Hospital /ID# 209273, Saga, Saga-ken
  - Tokitokai Tokito clinic /ID# 164218, Saitama-shi, Saitama
  - Shiga University of Medical Science Hospital /ID# 164323, Ōtsu, Shiga
  - Hamamatsu University Hospital /ID# 226729, Hamamatsu, Shizuoka
  - Matsuda Hospital - Hamamatsu /ID# 226831, Hamamatsu, Shizuoka
  - NHO Shizuoka Medical Center /ID# 164314, Sunto-gun, Shizuoka
  - Institute of Science Tokyo Hospital /ID# 164225, Bunkyo-ku, Tokyo
  - St. Lukes International Hospital /ID# 225969, Chuo-ku, Tokyo
  - Tokai University Hachioji Hospital /ID# 227102, Hachioji-shi, Tokyo
  - Kitasato University Kitasato Institute Hospital /ID# 164222, Minato-ku, Tokyo
  - Kyorin University Hospital /ID# 164226, Mitaka-shi, Tokyo
  - NTT Medical Center Tokyo /ID# 225595, Shinagawa-ku, Tokyo
  - Keio University Hospital /ID# 203630, Shinjuku-ku, Tokyo
  - Japanese Red Cross Wakayama Medical Center /ID# 171196, Wakayama, Wakayama
  - Wakayama Medical University Hospital /ID# 169485, Wakayama, Wakayama
  - Yamagata University Hospital /ID# 171481, Yamagata, Yamagata
  - Tokuyama Central Hospital /ID# 226857, Shunan-shi, Yamaguchi
  - The Jikei University Hospital /ID# 164279, Tokyo
  - Teikyo University Hospital /ID# 225594, Tokyo
- Latvia (2):
  - VCA Polyclinic Aura /ID# 160204, Riga
  - Pauls Stradins Clinical University Hospital /ID# 160205, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 201142, Kaunas
  - Vilnius University Hospital Santaros Klinikos /ID# 201144, Vilnius
- Mexico (3):
  - JM Research SC /ID# 206518, Cuernavaca, Morelos
  - Unidad de Atencion Medica e Investigacion en Salud /ID# 206515, Mérida, Yucatán
  - Health Pharma Professional Research S.A de C.V /ID# 206516, Del. Benito Juárez
- Netherlands (2):
  - Elisabeth Tweesteden Ziekenhuis /ID# 163738, Tilburg, North Brabant
  - Amsterdam UMC, locatie AMC /ID# 157965, Amsterdam, North Holland
- New Zealand (6):
  - Tauranga Hospital /ID# 212793, Tauranga South, Bay of Plenty
  - Christchurch Hospital. /ID# 205337, Christchurch, Canterbury
  - Dunedin Hospital /ID# 212791, Otago, Otago
  - Waikato Hospital /ID# 212788, Hamilton, Waikato Region
  - Hutt Hospital /ID# 212787, Lower Hutt, Wellington Region
  - Wellington Regional Hospital /ID# 205338, Newtown, Wellington Region
- Poland (12):
  - Vitamed Galaj i Cichomski Sp.j. /ID# 213358, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Gastromed Sp. z o.o /ID# 231065, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Plejady /ID# 170635, Krakow, Lesser Poland Voivodeship
  - Vistamed /ID# 210106, Wroclaw, Lower Silesian Voivodeship
  - Centrum Zdrowia MDM /ID# 170283, Warsaw, Masovian Voivodeship
  - Medical Network Sp.z.o.o. WIP Warsaw IBD Point Profesor Kierkus /ID# 216103, Warsaw, Masovian Voivodeship
  - Panstwowy Instytut Medyczny MSWiA w Warszawie /ID# 170286, Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sk?odowskiej-Curie Panstwowy Instytut Bada /ID# 170285, Warsaw, Masovian Voivodeship
  - Vivamed Sp. z o.o. /ID# 216308, Warsaw, Masovian Voivodeship
  - Endoskopia Sp. z o.o. /ID# 170284, Sopot, Pomeranian Voivodeship
  - NZOZ All-Medicus /ID# 170282, Katowice, Silesian Voivodeship
  - H-T Centrum Medyczne Endoterapia /ID# 231501, Tychy, Silesian Voivodeship
- Portugal (8):
  - Centro Hospitalar Do Alto Ave - Hospital Senhora Da Oliveira /ID# 165576, Guimarães, Braga District
  - Centro Hospitalar Universitário do Algarve, EPE - Hospital de Portimão /ID# 166563, Portimão, Faro District
  - Centro Hospitalar de Entre Douro e Vouga /ID# 166048, Santa Maria DA Feira, Porto District
  - Duplicate_Hospital Garcia de Orta, EPE /ID# 165579, Almada, Setúbal District
  - Unidade Local de Saude de Coimbra, EPE /ID# 166050, Coimbra
  - Duplicate_Centro Hospitalar Universitario Lisboa Central, EPE - Hospital dos Cap /ID# 165578, Lisbon
  - Unidade Local de Saude Sao Joao, EPE /ID# 165577, Porto
  - Centro Hosp de Tondela-Viseu /ID# 166049, Viseu
- Puerto Rico (2):
  - Ponce Medical School Foundation /ID# 222825, Ponce
  - VA Caribbean Healthcare System /ID# 222779, San Juan
- Romania (6):
  - Clinica Gastro Med SRL /ID# 224156, Cluj-Napoca, Cluj
  - Sana Monitoring /Id# 224154, Bucharest
  - Fundeni Clinical Institute /ID# 171259, Bucharest
  - Fundeni Clinical Institute /ID# 224155, Bucharest
  - Cabinet Particular Policlinic Algomed /ID# 171260, Timișoara
  - Duplicate_Centrul Medical Tuculanu SRL /ID# 171263, Timișoara
- Russia (17):
  - Interdisctrict Multidisciplinary Hospital /ID# 204921, Anzorey, Kabardino-Balkarskaya Respublika
  - GBUZ Allergology and Immunology Center of Ministry of Health of Kabardino-Bal /ID# 233974, Nal'chik, Kabardino-Balkarskaya Respublika
  - Immanuel Kant Baltic Federal University /ID# 204920, Kaliningrad, Kaliningrad Oblast
  - Kuzbass Regional Clinical Hospital /ID# 165759, Kemerovo, Kemerovo Oblast
  - Uninova Medical Center /ID# 229786, Saint Petersburg, Leningradskaya Oblast'
  - Arsvita Clinic /ID# 208947, Korolyov, Moscow Oblast
  - Novosibirski Gastrocenter /ID# 229852, Novosibirsk, Novosibirsk Oblast
  - Perm Clinical Center of the Federal Medical and Biological Agency /ID# 227456, Perm, Permskiy Kray
  - City Clinical Hospital #40 /ID# 204927, Sestroretsk, Sankt-Peterburg
  - Regional Clinical Hospital #1 /ID# 165763, Tyumen, Tyumen Oblast
  - Clinic of New Technologies of Medicine /ID# 204926, Dzerzhinskiy
  - First Moscow State Medical University n.a I.M. Sechenov /ID# 204981, Moscow
  - National Medical Research Center of Coloproctology n.a. A. N. Ryzhikh /ID# 203513, Moscow
  - Central Clinical Hospital RZHD Medicine /ID# 204922, Moscow
  - Euromedservice /ID# 204918, Pushkin
  - International Medical Center SOGAZ /ID# 206832, Saint Petersburg
  - Ulyanovsk Regional Clinical Hospital /ID# 204923, Ulyanovsk
- Serbia (6):
  - Clinical Hosp Center Zvezdara /ID# 200150, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 200153, Belgrade, Beograd
  - Clinical Hospital Center Dr Dragisa Misovic - Dedinje /ID# 224927, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 202060, Belgrade, Beograd
  - General Hospital Leskovac /ID# 224198, Leskovac, Jablanicki Okrug
  - Duplicate_Clinical Center Vojvodina /ID# 156876, Novi Sad, Vojvodina
- Mount Elizabeth Hospital /ID# 206563, Singapore, Central Singapore, Singapore
- Slovakia (4):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 164348, Banská Bystrica, Banská Bystrica Region
  - KM Management, spol. s.r.o. /ID# 206603, Nitra, Nitra Region
  - Fakultna nemocnica s poliklinikou Nove Zamky /ID# 224100, Nové Zámky, Nitra Region
  - Gastro I., s.r.o. /ID# 164345, Prešov, Presov
- Univ Medical Ctr Ljubljana /ID# 210628, Ljubljana, Slovenia
- South Africa (6):
  - Farmovs (Pty) Ltd /Id# 207538, Bloemfontein, Free State
  - Clinresco Centers /ID# 239825, Johannesburg, Gauteng
  - Allergy & Immunology (AIU) /ID# 171439, Cape Town, Western Cape
  - Dr JP Wright /ID# 171142, Cape Town, Western Cape
  - Private Practice Dr MN Rajabally /ID# 171141, Cape Town, Western Cape
  - Spoke Research Inc /ID# 229906, CAPE TOWN Milnerton, Western Cape
- South Korea (11):
  - Inje University Haeundae Hospital /ID# 203027, Busan, Busan Gwang Yeogsi
  - Dong-A University Medical Center /ID# 158665, Busan, Busan Gwang Yeogsi
  - Duplicate_Pusan National University Hospital /ID# 158670, Busan, Busan Gwang Yeogsi
  - The Catholic University of Korea, Daejeon St. Mary's Hospital /ID# 242379, Daejeon, Daejeon Gwang Yeogsi
  - Duplicate_Hanyang University Gurihospital /ID# 158661, Guri-si, Gyeonggido
  - CHA Bundang Medical Center /ID# 158669, Seongnam, Gyeonggido
  - The Catholic University Of Korea St. Vincent's Hospital /ID# 158664, Suwon, Gyeonggido
  - Kangbuk Samsung Hospital /ID# 158666, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 158663, Seoul, Seoul Teugbyeolsi
  - Yeungnam University Medical Center /ID# 158662, Daegu
  - Yonsei University Health System Severance Hospital /ID# 158660, Seoul
- Spain (12):
  - Hospital Arquitecto Marcide - Complejo Hospitalario Universitario de Ferrol /ID# 159463, Ferrol, A Coruna
  - Consorci Corporacio Sanitaria Parc Tauli Sabadell /ID# 159473, Sabadell, Barcelona
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 159466, Majadahonda, Madrid
  - Hospital Alvaro Cunqueiro CHUVI /ID# 167359, Vigo, Pontevedra
  - Hospital Universitario de Cabuenes /ID# 170745, Gijón, Principality of Asturias
  - Hospital Clinic de Barcelona /ID# 159462, Barcelona
  - Duplicate_Hospital Universitario Reina Sofia /ID# 167062, Córdoba
  - Hospital Universitario La Paz /ID# 159471, Madrid
  - Complejo Hospitalario Universitario de Pontevedra /ID# 216183, Pontevedra
  - Hospital Universitario de Salamanca /ID# 159469, Salamanca
  - Hospital Universitario Virgen Macarena /ID# 159969, Seville
  - Hospital Universitario Miguel Servet /ID# 159468, Zaragoza
- Sweden (3):
  - Alingsas lasarett /ID# 202075, Alingsås, Västra Götaland County
  - Sahlgrenska University Hospital Molndal /ID# 202841, Mölndal, Västra Götaland County
  - Danderyds sjukhus AB /ID# 202036, Stockholm
- Switzerland (2):
  - University Hospital Zurich /ID# 202908, Zurich, Canton of Zurich
  - Inselspital, Universitaetsspital Bern /ID# 202909, Bern
- Taiwan (6):
  - National Taiwan University Hospital /ID# 162188, Taipei City, Taipei
  - Chung Shan Medical University Hospital /ID# 171426, Taichung
  - China Medical University Hospital /ID# 160194, Taichung
  - Taichung Veterans General Hospital /ID# 171433, Taichung
  - Taipei Veterans General Hosp /ID# 171436, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 222878, Taoyuan
- Turkey (Türkiye) (9):
  - Acibadem Kozyatagi Hospital /ID# 213277, Kadıköy, Istanbul
  - Sisli Etfal Train & Res Hosp /ID# 171415, Şişli, Istanbul
  - Duplicate_Erciyes University Medical Fac /ID# 171283, Melikgazi, Kayseri
  - Ankara Univ Medical Faculty /ID# 167205, Ankara
  - Inonu Universitesi Turgut Ozal /ID# 203980, Battalgazi/malatya
  - Uludag University Medical Faculty /ID# 204179, Bursa
  - F?rat University Medical Facul /ID# 171285, Elâzığ
  - Istanbul Universitesi-Cerrahpasa Cerrahpasa Tip Fakultesi /ID# 167202, Istanbul
  - Duplicate_Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi /ID# 171290, Istanbul
- Ukraine (5):
  - CNE Regional Clinical Hospital of Ivano-Frankivsk RC /ID# 203366, Ivano-Frankivsk
  - Municipal Nonprofit Enterprise Kherson city clinical hospital n.a. Y.Y. Karabel /ID# 224349, Kherson
  - Medical Center OK Clinic LLC, International Institute of Clinical Research /ID# 205484, Kyiv
  - CNPE of Kyiv Regional Council Kyiv Regional Hospital /ID# 224344, Kyiv
  - Medical center of the private enterprise Sygma /ID# 224347, Kyiv
- United Kingdom (10):
  - Addenbrookes Hospital /ID# 158046, Cambridge, Cambridgeshire
  - Royal Devon & Exeter Hospital /ID# 157614, Exeter, Devon
  - Western General Hospital - NHS Lothian /ID# 208801, Edinburgh, Edinburgh, City of
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 157617, London, Greater London
  - Kings College Hospital NHS Foundation Trust /ID# 158762, London, Greater London
  - St George University Hospitals NHS Foundation Trust /ID# 208379, London, Greater London
  - University Hospital Southampton NHS Foundation Trust /ID# 210814, Southampton, Hampshire
  - Barnsley Hospital NHS Foundation Trust /ID# 202771, Barnsley
  - Liverpool University Hospitals NHS Foundation Trust /ID# 203860, Liverpool
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 158047, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Panaccione R, Melmed GY, Drobne D, Kaur M, Danese S, Hisamatsu T, Kalabic J, Chen S, Cheng L, Duan WR, Shah S, Louis E. Impact of Extended Risankizumab Treatment in Patients With Ulcerative Colitis Who Did Not Respond to Induction Treatment. Clin Gastroenterol Hepatol. 2025 Sep 13:S1542-3565(25)00797-9. doi: 10.1016/j.cgh.2025.09.007. Online ahead of print. PMID 40953785
- [Derived] Reinisch W, Loftus EV Jr, Schreiber S, Rubin DT, Louis E, Hecht PM, Barrachina EM, Kalabic J, Vladea R, Sharma D, Duan WR, Zhang Y, Panaccione R. Corticosteroid-sparing effects of risankizumab efficacy and safety in patients with moderately to severely active ulcerative colitis. J Crohns Colitis. 2025 Apr 4;19(4):jjaf025. doi: 10.1093/ecco-jcc/jjaf025. PMID 40168091
- [Derived] Panaccione R, Louis E, Colombel JF, D'Haens G, Peyrin-Biroulet L, Dubinsky M, Takeuchi K, Rubin DT, Kalabic J, Chien KB, Chen S, Cheng L, Zhang Y, Duan WR, Vladea R, Hecht PM, Morisset P, Schreiber S, Ferrante M. Risankizumab efficacy and safety based on prior inadequate response or intolerance to advanced therapy: post hoc analysis of the INSPIRE and COMMAND phase 3 studies. J Crohns Colitis. 2025 Jan 11;19(1):jjaf005. doi: 10.1093/ecco-jcc/jjaf005. PMID 39804294
- [Derived] Louis E, Schreiber S, Panaccione R, Bossuyt P, Biedermann L, Colombel JF, Parkes G, Peyrin-Biroulet L, D'Haens G, Hisamatsu T, Siegmund B, Wu K, Boland BS, Melmed GY, Armuzzi A, Levine P, Kalabic J, Chen S, Cheng L, Shu L, Duan WR, Pivorunas V, Sanchez Gonzalez Y, D'Cunha R, Neimark E, Wallace K, Atreya R, Ferrante M, Loftus EV Jr; INSPIRE and COMMAND Study Group. Risankizumab for Ulcerative Colitis: Two Randomized Clinical Trials. JAMA. 2024 Sep 17;332(11):881-897. doi: 10.1001/jama.2024.12414. PMID 39037800
- See also: Related Info. — https://www.abbvieclinicaltrials.com/study/?id=M16-066